CLINICAL TRIAL: NCT04479436
Title: A Multi-Center, Open-Label, Phase 2 Study to Evaluate Safety and Efficacy of U3-1402 in Subjects With Advanced or Metastatic Colorectal Cancer (CRC)
Brief Title: A Study to Evaluate U3-1402 in Subjects With Advanced or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early given the Interim Analysis for Part 1 (signal finding) did not meet pre-specified criteria and will not proceed to Part 2. Sponsor will proceed closing the study.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-U202; 2019-004418-32 (EudraCT Number)
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; U3-1402
MeSH Terms: conditions — Colorectal Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: HER3 High (IHC 3+, 2+) (Experimental): Cohort 1 participants will have high tumor expression levels of human epidermal receptor 3 (HER3) in a pre-treatment biopsy specimen.
  Interventions: Drug: Patritumab Deruxtecan
- Cohort 2: HER3 Low/Negative (IHC 1+, 0) (Experimental): Cohort 2 participants will have low or negative tumor expression levels of human epidermal receptor 3 (HER3) expression levels in a pre-treatment biopsy specimen.
  Interventions: Drug: Patritumab Deruxtecan

INTERVENTIONS:
Drug: Patritumab Deruxtecan — U3-1402 will be dosed at 5.6 mg/kg as an intravenous (IV) infusion administered on Day 1 of each 21-day cycle.
  Other Names: U3-1402

SUMMARY:
This study is designed to primarily evaluate the safety and efficacy of U3-1402 in participants with advanced or metastatic colorectal cancer (CRC) who have received at least 2 prior lines of therapy and will explore clinical benefit according to human epidermal growth factor receptor 3 (HER3) tumor expression level in otherwise refractory tumors.

DETAILED DESCRIPTION:
There will be 2 cohorts with enrollment in 2 parts. Participants will be treated on Day 1 of each 21-day cycle (every 3 weeks) with U3-1402 5.6 mg/kg intravenous (IV). The estimated treatment period is approximately 8 months and the follow-up period is approximately 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written informed consent prior to the start of any study specific procedures.
* Participants ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
* Pathological/histological confirmation of advanced or metastatic colon or rectal adenocarcinoma.
* Must be resistant, refractory, or intolerant to at least 2 prior lines of systemic therapy, that must include all of the following agents:

  * Fluoropyrimidine
  * Irinotecan
  * Platinum agents (e.g, oxaliplatin)
  * An anti-epidermal growth factor receptor (EGFR) agent, if clinically indicated
  * An anti-VEGF agent, if clinically indicated (eg, bevacizumab)
  * An immune checkpoint inhibitor (eg, microsatellite instability-high [MSI-H] status)
  * A BRAF inhibitor, if clinically indicated (eg, BRAF V600E positive)
* Has at least 1 measurable lesion confirmed by blinded independent central review (BICR) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1.
* Willing to provide a required pre-treatment tumor biopsy and an additional archival tissue sample for the assessment of HER3 expression levels by immunohistochemistry and exploratory biomarkers, defined as:

  1. Pre-treatment tumor biopsy. Participants may be exempted from the requirement to provide a pre-treatment tumor biopsy if archival tumor tissue was collected within 3 months of screening during or after treatment with the last prior cancer treatment and is of sufficient quantity (2 cores or 20 slides with adequate tumor tissue content).
  2. An additional archival tissue sample collected greater than 3 months prior to screening must be available and of sufficient quantity, as defined above, at the time of screening. If an archival tissue sample (collected greater than 3 months prior to screening) is not available, a subject may be included provided the pre-treatment tumor biopsy is obtained and after discussion and agreement from Sponsor (Medical Monitor or designee).
  3. Consent to provide on-treatment tumor biopsy. When at least 10 treatment tumor biopsies have been collected, the Sponsor will provide written notification of a change to the requirement.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Life expectancy ≥3 months.
* Has adequate bone marrow reserve and organ function at baseline based on local laboratory data defined as follows within 14 days prior to Cycle 1 Day 1:

  * Platelet count: ≥100,000/mm^3 or ≥100 × 10^9/L (platelet transfusions are not allowed up to 14 days prior to Cycle 1 Day 1 to meet eligibility)
  * Hemoglobin: ≥9.0 g/dL (transfusion and/or growth factor support is allowed)
  * Absolute neutrophil count: ≥1500/mm^3 or ≥1.5 × 10^9/L
  * Serum creatinine (SCr) OR creatinine clearance (CrCl): SCr ≤ 1.5 × upper limit of normal (ULN), OR CrCl ≥ 30 mL/min as calculated using the Cockcroft- Gault equation or measured CrCl; confirmation of CrCl is only required when creatinine is >1.5 × ULN
  * Alanine aminotransferase /aspartate aminotransferase: ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  * Total bilirubin: ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's syndrome [unconjugated hyperbilirubinemia] or liver metastases)
  * Serum albumin: ≥2.5 g/dL
  * Prothrombin time (PT) or PT-international normalized ratio (INR) and activated partial thromboplastin time (aPTT) / partial thromboplastin time (PTT): ≤1.5 × ULN except for subjects on coumarin- derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator

Exclusion Criteria:

* Any history of interstitial lung disease (including pulmonary fibrosis or radiation pneumonitis), has current interstitial lung disease (ILD), or is suspected to have such disease by imaging during screening.
* Clinically severe pulmonary compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  1. any underlying pulmonary disorder (e.g., pulmonary emboli, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion)
  2. any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis)

     * OR prior complete pneumonectomy.
* Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
* Evidence of leptomeningeal disease.
* Evidence of clinically active spinal cord compression or brain metastases
* Inadequate washout period prior to Cycle 1 Day 1 of U3-1402:

  1. Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days;
  2. Any cytotoxic chemotherapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study <14 days or 5 half-lives, whichever is longer;
  3. Monoclonal antibodies other than immune checkpoint inhibitors, such as bevacizumab (anti-VEGF) and cetuximab (anti-EGFRs) <28 days;
  4. Immune checkpoint inhibitor therapy <21 days;
  5. Major surgery (excluding placement of vascular access) <4 weeks;
  6. Radiotherapy treatment to >30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days;
  7. Chloroquine/hydroxychloroquine ≤14 days.
* Prior treatment with an anti-HER3 antibody and/or antibody drug conjugate (ADC) that consists of an exatecan derivative that is any topoisomerase I inhibitor (e.g, trastuzumab deruxtecan).
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 Grade ≤1 or baseline.
* Had primary malignancies other than CRC within 3 years prior to Cycle 1 Day 1, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated.
* Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day 1.
* Known Hepatitis B and/or Hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1.

  1. Participants with past or resolved hepatitis B virus (HBV) infection are eligible if:

     * Hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) positive; OR
     * HBsAg positive and HBV deoxyribonucleic acid (DNA) viral load is documented to be ≤2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases values (in the absence of liver metastasis); OR
     * HBsAg positive and HBV DNA viral load is documented to be ≤2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation for participants with liver metastasis and abnormal transaminases with a result of AST/ALT <3 × ULN.
  2. Participants with a history of hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (ie, sustained viral response according to the local product label but no less than 12 weeks, whichever is longer).
* Participant with any human immunodeficiency virus (HIV) infection.
* Any evidence of severe or uncontrolled systemic diseases (including active bleeding diatheses, active infection), psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the Investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (44):
- United States (21):
  - Highlands Oncology, Fayetteville, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation NMFF Hematology Oncology, Chicago, Illinois
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center University of Texas, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virgina Cancer Specialists, Fairfax, Virginia
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
- France (3):
  - Centre Georges-Franois Leclerc, Dijon
  - CHU Nantes, Nantes
  - Hospital St Antoine, Paris
- Asst Grande Ospedale Metropolitano Niguarda, Milan, Italy
- Japan (5):
  - Aichi Cancer Center Hospital, Nagoya, Nagoya-shi, Aichi-ken
  - National Hospital Organization - Osaka National Hospital (ONH), Osaka, Osaka-shi, Osaka-fu
  - Kindai University Hospital, Osaka, Osakasayama Shi
  - National Cancer Center Hospital East, Chiba
  - The Cancer Institute Hospital Of JFCR, Tokyo
- Poland (3):
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Ostrów Wielkopolski, Poznan
  - Szpital Kliniczny Przemienienia Pańskiego.University Hospital, Chemotherapy Department, Poznan
  - M Sklodowska Curie Memorial Cancer Center, Warsaw
- Spain (6):
  - Hospital del Mar - Institut Hospital del Mar d'Investigacions Mediques IMIM, Barcelona
  - VHIO Valle de Hebron Instituto de Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, CIOCC, Madrid
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (3):
  - Royal Marsden Hospital NHS, London
  - Sarah Cannon Research Institute UK, London
  - Sarah Cannon, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 12 sites. All 40 patients received at least one dose of study drug.
Groups:
- Cohort 1: HER3 High (IHC 3+, 2+): Participants in Cohort 1 had high tumor expression levels of human epidermal receptor 3 (HER3) and received an intravenous (IV) infusion of U3-1402 5.6 mg/kg on Day 1 of each 21-day cycle.
- Cohort 2: HER3 Low/Negative (IHC 1+, 0): Participants in Cohort 2 had low or negative tumor expression levels of human epidermal receptor 3 (HER3) expression levels and received an intravenous (IV) infusion of U3-1402 5.6 mg/kg on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+) | Cohort 2: HER3 Low/Negative (IHC 1+, 0)
Started | 39 | 1
Completed | 0 | 0
Not Completed | 39 | 1
Not completed — Progressive disease | 26 | 1
Not completed — Adverse Event | 6 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Clinical progression | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+) | Cohort 2: HER3 Low/Negative (IHC 1+, 0) | Total
Number analyzed (Participants) | 39 | 1 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 0 | 30
  >=65 years | 9 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — The mean age of Cohort 1 is being reported. Only 1 participant was enrolled in Cohort 2; the age of that participant is being reported.
  years | 57.0 (8.64) | 67 | 57.3 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 1 | 14
  Male | 26 | 0 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 26 | 1 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 1 | 30
  Japan | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) As Assessed By Blinded Independent Central Review (BICR) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: ORR defined as the proportion of participants with a best overall response of confirmed complete response (CR) or partial response (PR) as assessed by blinded independent central review. CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesion based on RECIST v1.1.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Overall response rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+) | Cohort 2: HER3 Low/Negative (IHC 1+, 0)
Number analyzed (Participants) | 39 | 1
Participants | 2 | 0

2. Secondary Outcome: Duration of Response (DoR) As Assessed by Blinded Independent Central Review (BICR) and Investigator Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: DoR defined as the time from the first documented response (CR or PR) to the date of disease progression or death due to any cause. CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions based on RECIST v1.1.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Duration of response was only assessed in patient responders in Cohort 1 of the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 2
months
  Duration of Response: BICR | 2.91 [2.79 to 3.02]
  Duration of Response: Investigator | 4.48 [2.56 to 6.41]

3. Secondary Outcome: Objective Response Rate (ORR) As Assessed by Investigator Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: ORR defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as assessed by Investigator. CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesion based on RECIST v1.1.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Objective response rate was assessed only in Cohort 1 of the Full Analysis Set. Per prespecified criteria cohort 2 was not able to be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
Participants | 2

4. Secondary Outcome: Disease Control Rate (DCR) by Blinded Independent Central Review (BICR) and Investigator Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: DCR is defined as the proportion of participants who achieved a confirmed best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD) as assessed by blinded independent central review or by the Investigator. Based on RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Disease control rate was assessed only in Cohort 1 of the Full Analysis Set. Per prespecified criteria cohort 2 was not able to be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
Participants
  Disease control rate (BICR) | 22
  Disease control rate (Investigator) | 22

5. Secondary Outcome: Time to Tumor Response (TTR) As Assessed by Blinded Independent Central Review (BICR) and Investigator Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: TTR defined as the time from the start of study treatment to the date of the first documentation of objective response (complete response [CR] or partial response [PR]) that is subsequently confirmed by Blinded Independent Central Review or by the Investigator. CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions based on RECIST v1.1.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Time to tumor response was assessed only in Cohort 1 responders who had a documented CR or PR in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 2
months
  Time to tumor response (BICR) | 1.99 (0.813)
  Time to tumor response (Investigator) | 1.53 (0.163)

6. Secondary Outcome: Progression-free Survival (PFS) Assessed by Blinded Independent Central Review (BICR) and Investigator Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: PFS is defined as the time from the start of study treatment to the date of the first documentation of objective PD or death due to any cause, whichever is earlier.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+) | Cohort 2: HER3 Low/Negative (IHC 1+, 0)
Number analyzed (Participants) | 39 | 1
months
  Progression-free survival (BICR) | 2.27 [1.51 to 2.96] | 5.5
  Progression-free survival (Investigator): number analyzed (Participants) | 39 | 0
  Progression-free survival (Investigator) | 2.53 [1.64 to 3.71] |

7. Secondary Outcome: Overall Survival (OS) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: OS defined as the time from the start of study treatment to the date of death due to any cause.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Overall survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+) | Cohort 2: HER3 Low/Negative (IHC 1+, 0)
Number analyzed (Participants) | 39 | 1
months | 10.58 [5.36 to 12.09] | 8.9

8. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Other Safety Parameters During the Study
Description: TEAEs, study-drug related TEAE, serious adverse events (SAE), study-drug related SAE, and adverse events of special interest (eg. interstitial lung disease and elevation of aminotransferases and total bilirubin) were assessed. A TEAE was defined as an AE with a start or worsening date during the on-treatment period. An SAE was an AE that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From Baseline (Day 0) to data cut off (up to approximately 16.5 months)
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: This cohort includes all patients with human epidermal receptor 3 (HER3) tumor expression (regardless of expression level) and received an intravenous (IV) infusion of U3-1402 5.6 mg/kg on Day 1 of each 21-day cycle.
Arm/Group | Overall
Number analyzed (Participants) | 40
Participants
  Treatment-emergent adverse events (TEAEs) | 40
  Study-drug related TEAE | 37
  Serious TEAE (SAE) | 17
  Study-drug related SAE | 9
  Adverse event of special interest (AESI) | 2

9. Secondary Outcome: Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline)
Description: Blood samples were collected to assess the immunogenicity of U3-1402.
Time Frame: At Baseline, and post-Baseline. Post-Baseline including any of the following timepoints- Cycle 1, Days 1&8; Cycles 2&4 and every 2 cycles thereafter, Day 1 (each cycle, 21 days), and at EOT (~16.5 months).
Population: Immunogenicity was assessed in the Safety Analysis Set only in Cohort 1. Per prespecified criteria cohort 2 was not able to be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
Participants
  Baseline: Positive | 0
  Baseline: Negative | 37
  Baseline: Missing | 2
  Post-baseline: Positive: number analyzed (Participants) | 38
  Post-baseline: Positive | 0
  Post-baseline: Negative: number analyzed (Participants) | 38
  Post-baseline: Negative | 38

10. Secondary Outcome: Number of Participants Who Have Treatment-emergent Anti-Drug Antibody (ADA)
Description: Blood samples were collected to assess the immunogenicity of U3-1402. Treatment-emergent ADA was defined as participants with a negative ADA status at Baseline who had a positive ADA status post-Baseline (treatment-induced ADA), or participants with a positive ADA status at both Baseline and post-Baseline but with an increase of at least 4-fold in ADA titer from Baseline to post-Baseline (treatment-boosted ADA), or participants who had missing ADA data at Baseline and had a positive ADA status post-Baseline.
Time Frame: as for outcome 9
Population: Immunogenicity was assessed in the Safety Analysis Set only in Cohort 1 participants at baseline and in participants post-baseline with at least 1 ADA sample. Per prespecified criteria cohort 2 was not able to be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
Participants
  Treatment-emergent ADA | 0
  Treatment-induced ADA | 0
  Treatment-boosted ADA | 0
  ADA missing at baseline but positive at post-baseline | 0

11. Secondary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter Cmax (antibody drug conjugate [ADC], total anti-HER3 antibody, and MAAA-1181a) were assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: At baseline (-8 hour to 0 hour), pre-infusion, and 15 minutes, 1 hour, 2 hour, 4 hour, and 8 hour post-infusion of Cycle 1 and Cycle 3 (each cycle is 21 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set only in Cohort 1 participants with available data. Per prespecified criteria cohort 2 was not able to be assessed
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
ug/mL
  U3-1402: Cycle 1 | 155.67 (43.45)
  U3-1402: Cycle 3: number analyzed (Participants) | 24
  U3-1402: Cycle 3 | 159.80 (47.94)
  Total anti-HER3 antibody: Cycle 1 | 154.08 (32.82)
  Total anti-HER3 antibody: Cycle 3: number analyzed (Participants) | 24
  Total anti-HER3 antibody: Cycle 3 | 153.86 (39.31)

12. Secondary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) of MAAA-1181a Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter Cmax of MAAA-1181a was assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
ng/mL
  Cycle 1 | 38.09 (19.68)
  Cycle 3: number analyzed (Participants) | 24
  Cycle 3 | 16.13 (9.29)

13. Secondary Outcome: Pharmacokinetic Parameter Time to Reach Maximum Serum Concentration (Tmax) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter Tmax (antibody drug conjugate [ADC], total anti-HER3 antibody, and MAAA-1181a) were assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 39
hours
  U3-1402: Cycle 1 | 2.42 [1.52 to 5.67]
  U3-1402: Cycle 3: number analyzed (Participants) | 24
  U3-1402: Cycle 3 | 4.39 [0.53 to 8.78]
  Total anti-HER3 antibody: Cycle 1 | 1.72 [1.45 to 505.50]
  Total anti-HER3 antibody: Cycle 3: number analyzed (Participants) | 24
  Total anti-HER3 antibody: Cycle 3 | 3.86 [0.53 to 8.78]
  MAAA-1181a: Cycle 1 | 5.28 [2.57 to 9.47]
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 24
  MAAA-1181a: Cycle 3 | 4.45 [0.65 to 8.33]

14. Secondary Outcome: Pharmacokinetic ParameterTrough Serum Concentration (Ctrough) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter Ctrough (antibody drug conjugate [ADC] and total anti-HER3 antibody) were assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: Pharmacokinetic paramters were assessed in the Pharmacokinetic Analysis Set only in Cohort 1 participants with available data. Per prespecified criteria cohort 2 was not able to be assessed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 35
ug/mL
  U3-1402: Cycle 1 | 7.98 (24.20)
  U3-1402: Cycle 3: number analyzed (Participants) | 15
  U3-1402: Cycle 3 | 12.76 (9.19)
  Total anti-HER3 antibody: Cycle 1 | 8.55 (29.61)
  Total anti-HER3 antibody: Cycle 3: number analyzed (Participants) | 15
  Total anti-HER3 antibody: Cycle 3 | 11.49 (9.25)

15. Secondary Outcome: Pharmacokinetic ParameterTrough Serum Concentration (Ctrough) of MAAA-1181a Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter Ctrough of MAAA-1181a was assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 35
ng/mL
  MAAA-1181a: Cycle 1 | 0.49 (1.42)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 16
  MAAA-1181a: Cycle 3 | 0.68 (0.66)

16. Secondary Outcome: Pharmacokinetic of Area Under the Serum Concentration-Time Curve Up to Last Quantifiable Time (AUClast) and During Dosing Interval (AUCtau) Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter AUC (antibody drug conjugate [ADC], total anti-HER3 antibody, and MAAA-1181a) were assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 20
day*ug/mL
  U3-1402, AUClast: Cycle 1 | 562.05 (246.93)
  U3-1402, AUClast: Cycle 3: number analyzed (Participants) | 0
  U3-1402, AUCtau: Cycle 1: number analyzed (Participants) | 18
  U3-1402, AUCtau: Cycle 1 | 569.42 (191.03)
  U3-1402, AUCtau: Cycle 3: number analyzed (Participants) | 7
  U3-1402, AUCtau: Cycle 3 | 1230.44 (257.08)
  Total anti-HER3 antibody, AUClast: Cycle 1 | 590.11 (279.67)
  Total anti-HER3 antibody, AUClast: Cycle 3: number analyzed (Participants) | 0
  Total anti-HER3 antibody, AUCtau: Cycle 1: number analyzed (Participants) | 18
  Total anti-HER3 antibody, AUCtau: Cycle 1 | 596.24 (217.23)
  Total anti-HER3 antibody, AUCtau: Cycle 3: number analyzed (Participants) | 9
  Total anti-HER3 antibody, AUCtau: Cycle 3 | 1104.22 (397.93)

17. Secondary Outcome: Pharmacokinetic of Area Under the Serum Concentration-Time Curve Up to Last Quantifiable Time (AUClast) and During Dosing Interval (AUCtau) of MAAA-1181a Following Administration of U3-1402 In Participants With Advanced or Metastatic Colorectal Cancer
Description: Serum PK parameter AUC of MAAA-1181a was assessed in the full PK sampling cohort using noncompartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Cohort 1: HER3 High (IHC 3+, 2+)
Number analyzed (Participants) | 20
day*ng/mL
  AUClast: Cycle 1 | 89.96 (60.43)
  AUClast: Cycle 3: number analyzed (Participants) | 0
  AUCtau: Cycle 1: number analyzed (Participants) | 17
  AUCtau: Cycle 1 | 92.81 (58.94)
  AUCtau: Cycle 3: number analyzed (Participants) | 5
  AUCtau: Cycle 3 | 78.68 (34.60)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for approximately 16.5 months.
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered pharmaceutical product and that does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  It was pre-specified that AE results would be presented for the overall subject population, rather than by cohort.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 23/40
Serious Adverse Events (participants affected / at risk) | 17/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=40)
Disease progression (General disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Nausea (General disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
International normalised ratio increased (Investigations) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Liver abscess (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pyelonephritis (Infections and infestations) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal obstruction (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=40)
Anaemia (Blood and lymphatic system disorders) | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 24
Oedema peripheral (General disorders) | 7
Pyrexia (General disorders) | 4
Disease progression (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 4
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 13
Lymphocyte count decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 17
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04479436/Prot_SAP_000.pdf